CLINICAL TRIAL: NCT01970618
Title: A Randomised, Double Blind, Placebo-controlled, Three Part Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Treatment With Single and Repeat Doses of Inhaled RV1162 in Healthy Subjects and Subjects With Chronic Obstructive Pulmonary Disease.
Brief Title: Safety, Tolerability and Pharmacokinetics (PK) of RV1162 in Healthy Subjects and COPD Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Respivert Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EST001; 2013 002329-44 (EudraCT Number)
Record Dates: First submitted 2013-10-22; First posted 2013-10-28 (Estimated); Last update posted 2014-11-20 (Estimated); Status verified 2014-11

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD); Healthy Volunteers
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Part A: single dose escalation (healthy subjects) (Experimental)
  Interventions: Drug: RV1162 single dose; Drug: RV1162 matching placebo single dose
- Part B: 7 day repeat dose (healthy subjects) (Experimental)
  Interventions: Drug: RV1162: 7 day repeat dose; Drug: RV1162 matching placebo: 7 day repeat dose
- Part C: 14 day repeat dose (COPD patients) (Experimental)
  Interventions: Drug: RV1162: 14 day repeat dose; Drug: RV1162 matching placebo: 14 day repeat dose

INTERVENTIONS:
Drug: RV1162 single dose — Safety and tolerability of single escalating doses
  Arms: Part A: single dose escalation (healthy subjects)
Drug: RV1162 matching placebo single dose — Safety and tolerability of single escalating doses
  Arms: Part A: single dose escalation (healthy subjects)
Drug: RV1162: 7 day repeat dose — Safety and tolerability of a repeat dose
  Arms: Part B: 7 day repeat dose (healthy subjects)
Drug: RV1162 matching placebo: 7 day repeat dose — Safety and tolerability of a repeat dose
  Arms: Part B: 7 day repeat dose (healthy subjects)
Drug: RV1162: 14 day repeat dose — Safety and tolerability of repeat escalating doses
  Arms: Part C: 14 day repeat dose (COPD patients)
Drug: RV1162 matching placebo: 14 day repeat dose — Safety and tolerability of repeat escalating doses
  Arms: Part C: 14 day repeat dose (COPD patients)

SUMMARY:
RV1162 is a new medicine being developed for possible treatment of smoking related lung disease (also known as chronic obstructive pulmonary disease - COPD). The main purpose of this study is to investigate the safety, tolerability and pharmacokinetics of single and repeat doses of RV1162.

ELIGIBILITY:
Inclusion Criteria (all subjects):

* Sign an informed consent document indicating they understand the purpose of and procedures required for the study and are willing to participate in the study.
* If a woman of childbearing potential, must have a documented menstrual period prior to the first dose and be willing and able to use 2 forms of contraception from screening until 4 months after the final dose of RV1162. Must not be a woman of child bearing potential for subjects in Part C, OR
* If a woman of non-childbearing potential must be amenorrhoeic for at least 1 year with an appropriate clinical profile, OR
* If a man, must be willing and able to use one of the contraception methods listed in the protocol and agree not to donate sperm, from the first dose until 4 months after the final dose of RV1162.
* Have a 12-lead ECG consistent with normal cardiac function
* Capable of complying with all study restrictions and procedures including ability to use the study inhaler correctly.

Parts A & B (healthy volunteers only)

* Aged between 18 and 50 years of age inclusive, at the time of signing the informed consent
* Healthy as determined by a physician, based on a full medical evaluation including medical history, physical examination and laboratory tests.
* Vital sign assessments within normal ranges
* Body mass index between 19 and 30 kg/m2 and body weight not less than 50 kg.
* Spirometry readings (FEV1 and FVC) to be ≥80% predicted value and FEV1/FVC ratio >0.7 at screening
* Are not taking prescription medications (with the exception of contraceptive or hormone replacement therapies) for 14 days prior to screening and agree not to use prescription medications throughout the duration of the study.
* Not taking over the counter medications for 14 days prior to screening and up to the final follow-up visit

Part C (COPD patients only)

* Aged between 40 and 75 years of age inclusive, at the time of signing the informed consent
* Have a diagnosis of COPD with symptoms compatible with COPD for at least 1 year
* COPD severity classification for GOLD Grade II/III
* Current or previous smoker with a smoking history of ≥ 10 pack years
* Not have a clinical abnormality or laboratory parameters outside the reference range
* Able to produce a viable induced sputum sample at the screening visit.

Exclusion Criteria (all subjects):

* Upper or lower respiratory tract infection within 4 weeks of screening
* Clinically significant abnormal values for haematology, clinical chemistry or urinalysis at screening
* History of, or a reason to believe a subject has a history of drug or alcohol abuse within the past 5 years
* Positive test for alcohol or drugs of abuse at screening or prior to dosing
* History of clinically significant allergies that would contraindicate participation
* Known allergy to the study drug or any of the excipients of the formulation
* Donated blood or blood products or had substantial loss of blood (more than 500 mL) within 3 months study drug or intention to donate blood or blood products during the study.
* Received an experimental drug or used an experimental medical device within 3 months or within a period less than 5 times the drug's half-life, whichever is longer, before the first dose of the study drug is scheduled.
* If a woman, has a positive pregnancy test at screening or admission, is pregnant, breast-feeding or planning to become pregnant during the study, or is a woman of child bearing potential (subjects in Part C).
* Positive test for human immunodeficiency virus (HIV) 1 and 2 antibodies, hepatitis B virus (HBV) infection, or hepatitis C antibodies.
* Preplanned surgery or procedures that would interfere with the conduct of the study.
* Employee of the Investigator or study centre, with direct involvement in the proposed study or other studies under the direction of that Investigator or study centre, as well as family members of the employees or the Investigator.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities
* History of regular alcohol consumption within 6 months of the study of an average weekly intake of >21 units for males, or >14 units for females
* The subject is unable or unwilling to comply fully with the study protocol
* Subject is mentally or legally incapacitated
* Unable or unwilling to undergo multiple venepuncture procedures or the subject has poor access to veins suitable for cannulation
* Any other reason that the Investigator considers makes the subject unsuitable to participate

Parts A & B (healthy volunteers only)

* History of smoking or use of nicotine-containing substances within the previous 6 months or a positive carbon monoxide test at screening or on admission

Part C (COPD patients only)

* A history of life-threatening COPD including Intensive Care Unit admission and/or requiring intubation
* A history of > 1 hospitalisation for COPD in the previous 2 years prior to screening
* Evidence of cor pulmonale or clinically significant pulmonary hypertension.
* Requires routine treatment for COPD using one of the restricted therapies listed in the protocol within the 6 weeks before screening
* A current diagnosis of asthma, active tuberculosis, lung cancer, bronchiectasis, sarcoidosis, lung fibrosis, interstitial lung diseases or other active pulmonary diseases
* A history of chronic uncontrolled diseases that the Investigator believes are clinically significant.
* A history of sleep apnoea.
* Previous lung resection or lung reduction surgery.
* Active participation in a pulmonary rehabilitation program
* Alanine transaminase (ALT) > 1.5 x upper limit of normal (ULN) at the screening visit.
* Major surgery, (requiring general anesthesia) within 6 weeks before the screening visit, or will not have fully recovered from surgery, or planned surgery through the end of the study
* A disclosed history, or one known to the Investigator, of significant noncompliance in previous investigational studies or with prescribed medications
* A history of unstable, or uncontrolled hypertension, or has been diagnosed with hypertension in last 3 months
* Any other reason that the Investigator considers makes the subject unsuitable to participate
* Vital sign assessments outside ranges: blood pressure between 100 and 160 mmHg systolic, inclusive, and between 55 and 100 mmHg diastolic; heart rate 50 - 100 bpm.
* Requires oxygen, even on an occasional basis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2013-10; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events | Cohorts 1 & 2, 42 days: Cohort 3, 15 days: Cohort 4, 21 days: Cohorts 5 & 6, 28 days,
  Assessment of the number of adverse events reported by subject following dosing
ECG assessment (12-lead ECG) | Cohorts 1 & 2, 42 days: Cohort 3, 15 days: Cohort 4, 21 days: Cohorts 5 & 6, 28 days
  Change from pre-dose values
Vital sign assessment (blood pressure and heart rate) | Cohorts 1 & 2, 42 days: Cohort 3, 15 days: Cohort 4, 21 days: Cohorts 5 & 6, 28 days
  Change from pre-dose values
Spirometry assessment (FEV1 & FVC) | Cohorts 1 & 2, 42 days: Cohort 3, 15 days: Cohort 4, 21 days: Cohorts 5 & 6, 28 days
  Change from pre-dose values
Clinical laboratory assessments (blood and urine samples) | Cohorts 1 & 2, 42 days: Cohort 3, 15 days: Cohort 4, 21 days: Cohorts 5 & 6, 28 days
  Change from pre-dose values

SECONDARY OUTCOMES:
Plasma RV1162 levels | Part A: Cohorts 1 & 2 x 4 treatment periods (TP), Cohort 3 x 1 TP (0, 10, 15 & 30 min, 1 ,2, 4, 6, 8, 10, 12 & 24h post-dose) each TP; Part B (Cohort 4): 34 samples up to 21 days post-dose; Part C (Cohorts 5 & 6): 46 samples up to 28 days post-dose
  Measurement of RV1162 in blood after dosing

OTHER OUTCOMES:
Serum biomarkers | Part C only: Day 1&14 (0,4&24h), Day 7 (0h), Day 28
  Measuring markers of inflammation in the blood
Exhaled breath condensate | Part C only: Screening, Days 1&14 (0&6h)
  Measuring markers of oxidative stress
Pulmonary plethysmography | Part C only: Admission, Day 14 (0h)
Sputum induction | Part C only: Screening, Day 12 and/or 14 (2h)
  To measure markers of inflammation in sputum

CONTACTS AND LOCATIONS:
Overall Officials: Jerome Boscia, MD, Study Director — Sponsor GmbH
Locations (1):
- Manchester, United Kingdom